CLINICAL TRIAL: NCT04678609
Title: Effects of Open and Closed Kinetic Chain Exercise on Functional Outcomes and Lower Limb Biomechanics in Mild Knee Osteoarthritis Patients
Brief Title: OKV Versus CKC for Biomechanics and Function in Mild Knee OA Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Shazlin Shaharudin, Lecturer, Universiti Sains Malaysia
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Supportive Care
Other Study IDs: USM/JEPeM/19100645
Record Dates: First submitted 2020-11-11; First posted 2020-12-22 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Osteoarthritis, Knee; Aging Problems
Keywords: biomechanics; exercise
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Open kinetic chain exercise (Experimental): In the OKC exercise group, participants will be taught by a physiotherapist about open kinetic chain exercises. Then, they will do the exercises at their home for eight weeks, with three session per week. The physiotherapist will contact the participants to monitor their adherence to the intervention. A diary is also provided to monitor their progress, pain level and any adverse events related to the intervention.
  Interventions: Other: Exercise
- Closed kinetic chain exercise (Experimental): In the OKC exercise group, participants will be taught by a physiotherapist about open kinetic chain exercises. Then, they will do the exercises at their home for eight weeks, with three session per week. The physiotherapist will contact the participants to monitor their adherence to the intervention. A diary is also provided to monitor their progress, pain level and any adverse events related to the intervention.
  Interventions: Other: Exercise
- Control (No Intervention): The untreated control group will receive patient's usual care of local government hospital which includes information about clinical manifestations, risk factors, diagnosis, treatment and nursing care for knee OA. Control group did not receive any home exercises guidance.

INTERVENTIONS:
Other: Exercise — CKC: exercise with joints fixed on the ground OKC: exercise with joints not fixed on the ground
  Arms: Closed kinetic chain exercise; Open kinetic chain exercise

SUMMARY:
Background: Clinical recommendations suggest exercises as the core treatment for knee osteoarthritis (OA) patients. However, the biomechanical modification following exercise therapy and its influence on pain remains unclear. The purpose of the study to compare the effectiveness of two different exercise programs, open kinetic chain (CKC) and closed kinetic chain (CKC) strengthening exercises, on pain and lower limb biomechanics for people more than 50 years old with painful mild grade knee OA.

Method: 66 individuals with mild knee OA, with knee pain in the previous one week, aged 50 years and above, and who have body mass index (BMI) between 18.9kg/m2 - 29.9 kg/m2 in Kelantan, Malaysia will be recruited in this study. Participants will be randomly allocated into three different groups, either OKC, CKC, or control groups. Participants in OKC and CKC groups will perform the exercises at their home three times per week for eight weeks. The control group will receive only the patient's clinical education about clinical manifestations, risk factors, diagnosis, treatment, and nursing care for knee OA and printed materials will be given. The outcome will be measured before and after the intervention. Primary outcomes are self-reported pain, disability, and quality of life scores. Secondary outcomes include lower limb biomechanics during gait and sit-to-stand, and knee isokinetic strength.

Discussion: This study will compare the efficacy of two different home-based exercise intervention programs for people with mild grade knee OA. Findings will provide valuable information for creating an effective exercise program that could slow down the progression of OA.

DETAILED DESCRIPTION:
The primary aim of this randomized controlled trial (RCT) is to compare the effects of two different home-based exercise programs namely OKC and CKC strengthening exercise intervention, on pain, disability, and quality of life on individuals with mild grade knee OA. Our secondary aim is to compare the effectiveness of OKC and CKC strengthening exercises on lower limb biomechanics during walking gait and sit to stand task. We hypothesize that after eight weeks of intervention OKC and CKC groups will show more improvements in pain, disability, and quality of life scores (what about the secondary outcomes) than the control group.

For the CKC and OKC exercise group, participants will perform an 8-week individualized home exercise, a minimum of three sessions in a week. Each session lasts about 30 minutes, including 5 minutes of walking as warming up session and quadriceps and hamstring stretching as the cooldown session. Daily Paracetamol 3000mg will be provided to all three groups. However, the consumption depends on each participant's needs, and the participants need to record it in the diary given. The exercise diary will be given to each participant to ensure patients' adherence to home exercise. During the intervention phase, a designated research team member will contact the participants personally to encourage them to continue their exercises.

The untreated control group received the patient's clinical education about clinical manifestations, risk factors, diagnosis, treatment, and nursing care for knee OA except the information related to exercise. The control group will not receive any home exercise guidance. Upon completing the trial, participants in the control group will receive either CKC or OKC exercises depending on their preference.

ELIGIBILITY:
Inclusion Criteria:

* female patients
* aged above 50
* body mass index (BMI) <30 kg / m2
* diagnosed with grade I and II knee OA using Kellgren-Lawrence
* have knee pain ≥ 2 on a VAS in the past week

Exclusion Criteria:

* have neurological disorders
* have implanted electrical devices
* have non-ambulatory status
* have significant cognitive impairment
* presence of systemic inflammatory arthritis
* have history of hip or knee arthroplasty
* have history of trauma or surgical arthroscopy of either knee in the last 6 months
* involved in a previous study that includes an exercise program within the last 6 months
* received a knee intra-articular injection within the last 3 months
* receives anticoagulant therapy
* have recent or imminent surgery within the last 3 months
* have any medical co-morbidities that excluding them from participation in exercises

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of pain intensity score at post-intervention | 8 weeks
  pain intensity will be assessed using a visual analogue scale. It consists of a bidirectional 10-cm straight line, where 0 cm is "no pain" and 10 cm is "worst imaginable pain," located at either end of the line. Patients will be instructed to draw a vertical mark on the line indicating their pain level.
Change from baseline of disability score at post-intervention | 8 weeks
  Western Ontario and McMaster Universities Arthritis Index consists of a number of questions designed to assess the clinical severity of the disease (5 questions for pain, 2 questions for stiffness and 17 questions for physical function). It includes 24 questions, each question scored using a five-point scale (0-4) with higher scores representing greater levels of pain, stiffness and severity of the disease. The overall score (index) is determined by summing the scores across the three dimensions and the score ranges between 0-96 (derived from a 0-4 Likert scale).
Change from baseline of quality of life score at post-intervention | 8 weeks
  The Osteoarthritis Knee and Hip Quality of Life in Malay Version consists of 43 items divided into five dimensions: physical activity, mental health, pain, social support, and social functioning Each item in the five dimensions is measured on a numerical rating scale from 0 to 10. Each item is scored on a scale from 0 to 10, and the normalized scores were obtained by computing the sum of item scores for each domain and calculated to a scale from 0 (worst) to 100 (best) possible quality of life.

SECONDARY OUTCOMES:
Change from baseline of speed during gait at post-intervention | 8 weeks
  The time taken to complete a 6 metre platform will be determined before and after intervention. Faster speed indicates improve function.
Change from baseline of knee adduction moment during gait at post-intervention | 8 weeks
  The knee adduction moment calculated from the vertical ground reaction force will be collected during mid-stance phase of gait. The value is in Newton metre and will be compared pre- and post-intervention. Reduced knee adduction moment indicates improved biomechanics.

CONTACTS AND LOCATIONS:
Overall Officials: Shazlin Shaharudin, PhD, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- Universiti Sains Malaysia, Kota Bharu, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No
All forms are anonymous and will be entered into SPSS software. Only research team members can access the data. Data will be presented as grouped data and will not identify the responders individually.

REFERENCES:
- [Derived] Ng WH, Jamaludin NI, Sahabuddin FNA, Ab Rahman S, Ahmed Shokri A, Shaharudin S. Comparison of the open kinetic chain and closed kinetic chain strengthening exercises on pain perception and lower limb biomechanics of patients with mild knee osteoarthritis: a randomized controlled trial protocol. Trials. 2022 Apr 15;23(1):315. doi: 10.1186/s13063-022-06153-8. PMID 35428274